CLINICAL TRIAL: NCT05631899
Title: A Pilot Clinical Trial of Autologous EphA-2-Targeting Chimeric Antigen Receptor Dendritic Cell Vaccine Loaded With KRAS Mutant Peptide in Combination With Anti-PD-1 Antibody/Anti-CTLA4 Antibody for Local Advanced/Metastatic Solid Tumors.
Brief Title: CAR-DC Vaccine and ICIs in Local Advanced/Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-074
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor, Adult; EphA2 Overexpression; KRAS G12V; KRAS G12C; KRAS G12D
Keywords: Local Advanced/Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel; Cyclophosphamide; Injections; spartalizumab; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KRAS-EphA-2-CAR-DC (Experimental): In the priming phase, a conditioning chemotherapy regimen of Abraxane and cyclophosphamide is administered three days before vaccination, and KRAS-EphA-2-CAR-DC vaccine is infused on Day 0 and Day 7 in Week 1.
  In the boost phase, KRAS-EphA-2-CAR-DC vaccine is infused one dose every 4 weeks since Week 5 for a total of 6 to 8 doses, then maintenance vaccination is given one dose every 8 weeks, until:
  1. Unacceptable toxicity occurred or disease progression; or
  2. Reactive T cells are undetected repeatedly after the last vaccine dose; or
  3. Vaccine exhaustion.
  Interventions: Biological: KRAS-EphA-2-CAR-DC; Drug: Abraxane; Drug: Cyclophosphamide
- KRAS-EphA-2-CAR-DC plus anti-PD-1 antibody (Experimental): In the priming phase, a conditioning chemotherapy regimen of Abraxane and cyclophosphamide is administered three days before vaccination, and KRAS-EphA-2-CAR-DC vaccine is infused on Day 0 and Day 7 in Week 1.
  In the boost phase, KRAS-EphA-2-CAR-DC vaccine is infused one dose every 4 weeks since Week 5 for a total of 6 to 8 doses, then maintenance vaccination is given one dose every 8 weeks.
  Anti-PD-1 antibody is administered 2 days after the first dose of KRAS-EphA-2-CAR-DC vaccine in the boost phase (Day 3 in Week 5) and every 4 weeks afterwards, until:
  1. Unacceptable toxicity occurred or disease progression; or
  2. Reactive T cells are undetected repeatedly after the last vaccine dose; or
  3. Vaccine exhaustion.
  Interventions: Biological: KRAS-EphA-2-CAR-DC; Drug: Abraxane; Drug: Cyclophosphamide; Drug: Anti-PD-1 antibody
- KRAS-EphA-2-CAR-DC plus anti-PD-1 antibody and anti-CTLA4 antibody (Experimental): In the priming phase, a conditioning chemotherapy regimen of Abraxane and cyclophosphamide is administered three days before vaccination, and KRAS-EphA-2-CAR-DC vaccine is infused on Day 0 and Day 7 in Week 1.
  In the boost phase, KRAS-EphA-2-CAR-DC vaccine is infused one dose every 8 weeks since Week 5.
  Anti-PD-1 antibody and anti-CTLA4 antibody are administered 2 days after the first dose of KRAS-EphA-2-CAR-DC vaccine in the boost phase (Day 3 in Week 5) and every 3 weeks afterwards for four doses, followed by anti-PD-1 antibody once every 3 weeks, until:
  1. Unacceptable toxicity occurred or disease progression; or
  2. Reactive T cells are undetected repeatedly after the last vaccine dose; or
  3. Vaccine exhaustion.
  Interventions: Biological: KRAS-EphA-2-CAR-DC; Drug: Abraxane; Drug: Cyclophosphamide; Drug: Anti-PD-1 antibody; Drug: Anti-CTLA4 Monoclonal Antibody

INTERVENTIONS:
Biological: KRAS-EphA-2-CAR-DC — 5~10 × 10^6 CAR-DCs per dose will be administered by intravenous injection.
Drug: Abraxane — Intravenous abraxane 125 mg/m^2/day on day-5.
  Other Names: Abraxane Injectable Product
Drug: Cyclophosphamide — Intravenous cyclophosphamide 300 mg/m^2/day on day -4.
  Other Names: Cyclophosphamide for Injection
Drug: Anti-PD-1 antibody — Intravenous anti-PD-1 antibody 200 mg/day.
  Other Names: PD-1 blocking antibody
  Arms: KRAS-EphA-2-CAR-DC plus anti-PD-1 antibody; KRAS-EphA-2-CAR-DC plus anti-PD-1 antibody and anti-CTLA4 antibody
Drug: Anti-CTLA4 Monoclonal Antibody — Intravenous anti-CTLA4 antibody 1 mg/kg/day
  Other Names: Ipilimumab
  Arms: KRAS-EphA-2-CAR-DC plus anti-PD-1 antibody and anti-CTLA4 antibody

SUMMARY:
This is a pilot clinical trial for subjects with local advanced/metastatic solid tumors to determine the safety, efficacy and immune response of autologous EphA2-targeting CAR-DC vaccine loaded with KRAS mutant peptide (KRAS-EphA-2-CAR-DC) in combination with ICIs. It aims to: assess the safety and antitumor effects of KRAS-EphA-2-CAR-DC vaccine; detect T cell response against KRAS mutant peptide and tumor neoepitopes after the treatment with KRAS-EphA-2-CAR-DC vaccine and ICIs.

DETAILED DESCRIPTION:
Therapeutic cancer vaccines, especially DC-based vaccines, are extensively pursued immune approaches in addition to immune checkpoint blockade antibodies and chimeric antigen receptor T cells. DCs can engulf, process and present tumor antigens to T cells, thereby initiating a potent and tumor-specific immune response. However, clinical outcomes of therapeutic cancer vaccines still remain poor, with objective response rates that rarely exceed ~15%. The maturation and activation of DCs are necessary steps to trigger the antitumor responses. However, it is increasingly clear that tumor-infiltrating dendritic cells (TIDCs) usually have an immature or tolerated phenotype that plays central roles in developing tumor microenvironment (TME). As a consequence, malfunction of TIDCs could suppress the infiltration and function of tumor infiltrating T cells and convert them into immune suppressive regulatory T cells.

In our previous research, we constructed novel CAR-DCs (Chimeric antigen receptor engineered dendritic cells) containing a scFv domain targeting EphA2 antigen, CD8a transmembrane, tandem DC-specific activation domains. The engineered CAR-DCs were activated when contacting with tumor targets in TME, and consequently, augmented the cytotoxicity of antigen specific T cells in immune system humanized solid tumor mouse models. Our design of CAR-DCs provides an effective vaccine strategy for solid tumors. Therefore, we designed an autologous CAR-DC vaccine engineered with anti-EphA2 CAR and KRAS mutant peptide (KRAS-EphA-2-CAR-DC) , which can suppress the growth of tumors expressing the correlated KRAS mutant in animal models. In addition, the combination of the immune checkpoint inhibitors could further reverse immunosuppressive TME and globally activate T cell responses. In this pilot study, we aim to assess the safety, efficacy and immune response of KRAS-EphA-2-CAR-DC combined with anti-PD-1 antibody/anti-CTLA4 antibody in patients with local advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. ECOG performance status ≤2 and Estimated life expectancy of more than 3 months.
3. Local advanced/metastatic solid tumors confirmed by histopathology or cytology with documentation of tumor EphA2 positive (≥20%) and KRAS mutation (G12V or G12D or G12C) within 6 months prior to screening. The second malignancy is allowed.
4. No clinical response to standard frontline therapy, or no standard therapy exists. Patients who have declined standard therapy or have no access to standard therapy may be enrolled and the reasons for lack of access need to be documented. Previous treatment with anti-PD-1/PD-L1 antibodies or anti-CTLA4 antibody are allowed, regardless of the level of PD-1/PD-L1 expression, dMMR and TMB.
5. At least one measurable lesion at baseline per RECIST version 1.1.
6. Adequate organ function as defined by the following criteria: ANC ≥1000 cells/μL; Platelet count ≥80,000/μL; Hemoglobin ≥8.0 g/dL; Serum AST and serum ALT, ≤3.0 x ULN (≤5 x ULN for patients with liver metastases); Total serum bilirubin ≤3.0 x ULN); Serum creatinine ≤2 x ULN or creatinine clearance of ≥45 mL/min.
7. Willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
8. Willing to complete all scheduled visits and assessments at the institution administering therapy.
9. Able to read, understand and provide written informed consent.

Exclusion Criteria:

1. Having KRAS (G12V or G12D or G12C) germline mutation.
2. Active central nervous system disease involvement (but allow patients with prior brain metastases treated at least 4 weeks prior to enrollment that are clinically stable and do not require intervention), or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity.
3. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation.
4. Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
5. Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS).
6. Active infection of hepatitis B virus (HBV), or hepatitis C virus (HCV).
7. Patients with history (within the last 5 years) or risk of autoimmune disease who have immunosuppressive medications or immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone or equivalent) within 28 days prior to enrollment. However, patients who received a short course of corticosteroids (eg, premedication prior to antibody drug) will be eligible for study entry.
8. Major trauma or major surgery within 4 weeks prior to enrollment.
9. Previous treatment involving KRAS mutant (G12V or G12D or G12C) and EphA2.
10. Systemic chemotherapy and other intervene within 2 weeks prior to vaccination.
11. Being participating or withdrew any other trials within 4 weeks.
12. Any serious underlying medical (eg, pulmonary, renal, hepatic, gastrointestinal, or neurological) or psychiatric condition or any issue that would limit compliance with study requirements.
13. Vaccination within 30 days of study enrollment.
14. Pregnant, lactating, or breastfeeding females.
15. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events (AEs) | 2 years
  Determining the safety profile following the initiation of treatment and grading these toxicities by CTCAE v5.0. AEs such as cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Clinical Response | 2 years
  Clinical response will be determined by RECIST 1.1 and iRECIST criteria. Response rate is the proportion of patients that achieve CR and PR.
Disease Control | 2 years
  Disease control will be determined by RECIST 1.1 and iRECIST criteria. Disease control rate is the proportion of patients that achieve CR, PR and SD.
Immune Response | Peripheral blood: baseline, weekly before Week 9, prior to each vaccination after Week 9 until last vaccination and 1 year after last vaccine. Tumor tissue: baseline, Week 3, and following timing will be performed according to subject's condition.
  Immune response will be evaluated by phenotype and functional analysis of vaccine-reactive T cells and Neoantigen-reactive T cells as well as other immune cells in peripheral blood and tumor samples. Response is defined by ≥3 folds increase relative to pre-vaccination.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from KRAS-EphA-2-CAR-DCs infusion to documented disease progression or death.
Overall Survival (OS) | 2 years
  OS is defined as the time from KRAS-EphA-2-CAR-DCs infusion to the date of death.
Time to response (TTR) | 2 years
  TTR is defined as the time from KRAS-EphA-2-CAR-DCs infusion to first assessed CR or PR by investigators and based on the iRECIST criteria.
Duration of response (DOR) | 2 years
  DOR is defined as the time from objective response (OR) until documented tumor progression date among responders.
Number and copy number of KRAS-EphA-2-CAR-DCs | Peripheral blood samples are collected on days 0, 3, 7, 10, 22, the day before each vaccination until last vaccination and 1 year after last vaccine. Tumor tissues are collected at baseline, the day before Week 5, and after combination.
  Number and copy number of KRAS-EphA-2-CAR-DCs were assessed by number in peripheral blood and tumor tissue.
The level of cytokines in serum | Peripheral blood samples are collected on days 0, 3, 7, 10, 22, the days before each vaccination until last vaccination and 1 year after last vaccine. Tumor tissues are collected at baseline, the day before Week 5, and after combination.
  The cytokines mainly include IL-1, IL-2, IL-6, IL-8, IL-10, IL-12 (p70), TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, Ph.D, Study Director — Zhejiang University
Locations (1):
- Biotherapeutic Department of Chinsese PLA Gereral Hospital, Beijing, Beijing Municipality, China